CLINICAL TRIAL: NCT00590499
Title: A Prospective Survey of Emergent Agitation Following Craniotomy: Incidence, Risk Factors and Outcomes
Brief Title: Agitation in Post Operative Neurosurgical Patients
Status: Completed | Type: Observational
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Jian-Xin Zhou, Professor, Capital Medical University
Other Study IDs: BJTTH-ICU-07-012
Record Dates: First submitted 2007-12-26; First posted 2008-01-10 (Estimated); Last update posted 2014-01-31 (Estimated); Status verified 2014-01

CONDITIONS: Agitation; Craniotomy
Keywords: agitation; craniotomy; incidence; risk factor; outcome
MeSH Terms: conditions — Psychomotor Agitation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- agitation group: The Riker sedation-agitated scale (SAS) levels 5-7.
- non-agitation group: The Riker sedation-agitated scale (SAS) levels 1-4.

SUMMARY:
Agitation is a significant clinical issue in anesthesiology and critical care medicine. Several studies have carried out to survey the epidemics of agitation in post-anesthesia care unit and intensive care unit, and results revealed that agitation had an adverse impact on outcomes. To our clinical experience, agitation can occur in postoperative neurosurgical patients, and is often difficult to manage. However, agitation in this subset of patients is poorly evaluated. In present study, adult patients following craniotomy will be enrolled consecutively, and incidence, risk factor and outcome of emergent agitation will be investigated. The results of the study will provide basic data for prevention and treatment of agitation in postoperative neurosurgical patients.

DETAILED DESCRIPTION:
The study will enroll 120 consecutive adult patients admitted to Neuro-ICU for post-operative care following craniotomy. Sedation-Agitation Scale (SAS) will be evaluated and documented every hour or as needed during stay in ICU by nurse on duty. Emergent agitation is defined as SAS of 5 to 7 at anytime during the first 24 hr of ICU stay.Patients are divided into 2 groups: non-agitation group (SAS 1-4) and agitation group (SAS 5-7).Data collection includes pre-operative records, events during anesthesia and operation, events during ICU stay, and outcomes. The primary outcome is complications such as self-removal of endotracheal tube, central venous or bladder catheters. The secondary and third outcomes are ICU stay and Glasgow Outcome Scale at hospital discharge, respectively. Incidence of agitation will be calculated to present an epidemiological knowledge. Univariate analyses between the two groups will be used for preliminary selection of model variables. Then stepwise block logistic regression will be applied to model the risk of agitation using significant univariate predictors.

ELIGIBILITY:
Inclusion Criteria:

* adult patients admitted to Neuro-ICU for post-operative care following craniotomy

Exclusion Criteria:

* age<18 yr old
* time interval between operation to ICU admission is longer than 24 hr
* re-operation within 72 hr
* persistently comatose during first 24 hr after operation (GCS≤8)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 120 consecutive adult patients admitted to Neuro-ICU for post-operative care following craniotomy
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2012-07; Primary Completion 2012-12 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Complications: self-removal of endotracheal tube, central venous or bladder catheters. | 24 hours

SECONDARY OUTCOMES:
ICU stay and Glasgow Outcome Scale | At hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Jian-Xin Zhou, MD, Study Chair — ICU, Beijing Tiantan Hospital
Locations (1):
- Jian-Xin Zhou, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Chen L, Xu M, Li GY, Cai WX, Zhou JX. Incidence, Risk Factors and Consequences of Emergence Agitation in Adult Patients after Elective Craniotomy for Brain Tumor: A Prospective Cohort Study. PLoS One. 2014 Dec 10;9(12):e114239. doi: 10.1371/journal.pone.0114239. eCollection 2014. PMID 25493435